CLINICAL TRIAL: NCT07301645
Title: Efficacy of 3D Versus 2D Movie Viewing on Stereopsis and Visual Function in Children With Residual Ambliopia. A Randomized Controlled Trial.
Brief Title: VISION-3D: Visual Skills Improvement With On-screen 3D Movies.
Acronym: VISION3D
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Politècnica de Catalunya (Other)
Collaborators: Hospital Universitari Mutua Terrassa (Unknown)
Responsible Party: Principal Investigator, Laura Asensio Jurado, Principal Investigator, Universitat Politècnica de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDE1LAJ.VISION3D
Record Dates: First submitted 2025-11-26; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Amblyopia; Strabismus
Keywords: Amblyopia; Strabismus; Cinema 3D
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Intervention Model Description: Randomized parallel-group with delayed-treatment (wait-list) extension.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Movie Viewing (Experimental)
  Interventions: Behavioral: Stereoscopic (3D) Movie Viewing
- 2D Movie Viewing (Active Comparator)
  Interventions: Behavioral: 2D Movie Viewing

INTERVENTIONS:
Behavioral: Stereoscopic (3D) Movie Viewing — Repeated binocular visual stimulation. Participants view age-appropriate commercial films under standardized conditions once a week for three consecutive weeks in Phase 1. In the experimental intervention, the films are viewed in stereoscopic 3D using active shutter glasses and a calibrated 3D projection system. Each session lasts 90-120 minutes. After Phase 1, all participants receive three additional weekly 3D sessions (delayed treatment extension).
  Arms: 3D Movie Viewing
Behavioral: 2D Movie Viewing — Repeated binocular visual stimulation. Participants view age-appropriate commercial films under standardized conditions once a week for three consecutive weeks in Phase 1. In the control intervention, the films are viewed in 2D with identical duration and setting. Each session lasts 90-120 minutes. After Phase 1, all participants receive three additional weekly 3D sessions (delayed treatment extension).
  Arms: 2D Movie Viewing

SUMMARY:
This clinical study investigates whether watching 3D films can help improve the vision of children with residual amblyopia (lazy eye), that is, those children who, despite having undergone usual treatments such as glasses or patching, still maintain some visual deficit. The main objective is to verify whether viewing in 3D is better than viewing in 2D in improving depth vision (stereopsis), visual acuity and ocular alignment. The hypothesis is that 3D films, by providing richer binocular stimuli, will produce greater improvements than the same 2D films.

Children between 4 and 14 years of age with residual, stable and previously treated unilateral amblyopia will be included. Participants will be recruited from the pediatric ophthalmology/optometry clinics of the Mútua University Hospital

The study will be conducted in two locations: the visual examinations will be performed at the Mútua University Hospital in Terrassa, and the film sessions at the Faculty of Optics and Optometry of Terrassa (FOOT, UPC), in rooms prepared with a projector and 3D glasses.

The design is randomized and controlled. In a first phase, the children will be randomly divided into two groups: one group will watch 3 films in 3D and the other will watch the same films in 2D. Then, in a second phase, all participants will watch 3 additional sessions in 3D. Four evaluation visits will be made: before starting, after phase 1, after phase 2 and a follow-up two months later. These visits will measure stereopsis, visual acuity, and ocular deviation with standard optometric tests.

Watching 3D movies is a safe and non-invasive activity; therefore, no significant risks are expected beyond some possible mild and transient discomfort such as eye strain or headache, which will be recorded if it occurs. Potential benefits include improved depth perception and other visual functions, and the results could open the door to new, fun and motivating therapeutic options for other children with amblyopia in the future.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 12 years.
* Previous diagnosis of unilateral amblyopia (anisometropic, strabismic, or mixed).
* History of conventional treatment (optical correction, occlusion and/or penalization) with stable visual acuity for at least 6 months.
* Interocular visual acuity difference ≥ 0.2 logMAR (≈ ≥2 Snellen lines).
* Ability to understand and follow age-appropriate basic instructions.
* Parent/guardian consent (and child assent when applicable)

Exclusion Criteria:

* Ocular surgery within the last 6 months.
* Manifest strabismus >15 prism diopters.
* Concomitant ocular pathology that may affect vision (e.g., cataract, nystagmus, ptosis, corneal opacity, retinal disease, optic neuropathy).
* Cognitive or neurological deficits preventing compliance with the protocol.
* Prior intensive exposure to 3D cinema or VR/3D videogames that could act as a confounder.
* Family or child refusal to participate

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in stereoacuity measured with the Random Dot 2 Stereo Test (log arcsec) | Baseline (T0, Week 0), post-Phase 1 (T1, Week 3), post-Phase 2 (T2, Week 6), and follow-up (T3, 2 months after Phase 2)
  Stereoacuity will be assessed using the validated Random Dot 2 Stereo Test. Results will be recorded in arcseconds and analyzed as log arcsec. The primary endpoint is the change from baseline (T0) to each post-intervention assessment (T1 and T2) and follow-up (T3).
Change from baseline in best-corrected visual acuity (BCVA) of the amblyopic eye measured with ETDRS (logMAR) | Baseline (T0, Week 0), post-Phase 1 (T1, Week 3), post-Phase 2 (T2, Week 6), and follow-up (T3, 2 months after Phase 2).
  Best-corrected visual acuity of the amblyopic eye will be assessed using standardized ETDRS optotypes with the participant wearing habitual optical correction. Visual acuity will be recorded in logMAR. The outcome is the change in BCVA from baseline (T0) to each post-intervention assessment (T1 and T2) and follow-up (T3).
Change from baseline in ocular deviation measured by cover test with prism bars at distance (6 m) and near (40 cm) (prism diopters) | Baseline (T0, Week 0), post-Phase 1 (T1, Week 3), post-Phase 2 (T2, Week 6), and follow-up (T3, 2 months after Phase 2)
  Ocular deviation will be assessed using the cover test with prism bars at distance (6 m) and near (40 cm). The magnitude and direction of deviation will be recorded in prism diopters (PD/DP), distinguishing esotropia and exotropia when present. The outcome is the change in ocular deviation from baseline (T0) to each post-intervention assessment (T1 and T2) and follow-up (T3).

SECONDARY OUTCOMES:
Change from baseline in binocular sensory status (suppression/fusion) measured by the Worth 4 Dot test at distance and near. | Baseline (T0, Week 0), post-Phase 1 (T1, Week 3), post-Phase 2 (T2, Week 6), and follow-up (T3, 2 months after Phase 2).
  Binocular sensory status will be assessed using the Worth 4 Dot test at distance and near. Participants will be classified as showing fusion or suppression (and, if applicable, diplopia) based on standard Worth 4 Dot criteria. The outcome is the change in binocular sensory status from baseline (T0) to post-intervention assessments (T1 and T2) and follow-up (T3).
Retinal correspondence status assessed by the Bagolini striated lens test | Baseline (T0, Week 0), post-Phase 1 (T1, Week 3), post-Phase 2 (T2, Week 6), and follow-up (T3, 2 months after Phase 2)
  Retinal correspondence will be evaluated using the Bagolini striated lens test under standard clinical conditions. Participants will be classified as showing normal retinal correspondence, anomalous retinal correspondence, or suppression according to Bagolini response patterns. Results will be reported at each assessment time point.
Vision-related quality of life measured by the Pediatric Eye Questionnaire (PedEyeQ) total score | Baseline (T0, Week 0), post-Phase 1 (T1, Week 3), post-Phase 2 (T2, Week 6).
  Vision-related quality of life will be assessed using the age-appropriate PedEyeQ modules (child self-report and/or parent-proxy, plus parent component). Total PedEyeQ scores will be calculated according to the scoring manual and reported at each assessment time point.
Participant/family satisfaction with the intervention measured by a study-specific Likert satisfaction questionnaire | Post-Phase 1 (T1, Week 3), post-Phase 2 (T2, Week 6).
  Participant/family satisfaction will be measured using a structured study-specific questionnaire with Likert-type items (e.g., enjoyment, comfort, perceived benefit, and willingness to repeat). Satisfaction scores will be summarized and reported by group at each post-intervention time point.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mohan V. Dietary fibre and ischaemic heart disease. J Assoc Physicians India. 2000 Sep;48(9):869-70. No abstract available. PMID 11198783